CLINICAL TRIAL: NCT01012609
Title: A Phase II Trial of External Beam Radiation Therapy and Cetuximab Followed by Irinotecan and Cetuximab for Children and Young Adults With Newly Diagnosed Diffuse Pontine Tumors and High-Grade Astrocytomas (POE08-01)
Brief Title: External Beam Radiation Therapy and Cetuximab Followed by Irinotecan and Cetuximab for Children and Young Adults With Newly Diagnosed Diffuse Pontine Tumors and High-Grade Astrocytomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Children's Healthcare of Atlanta (Other); Dana-Farber Cancer Institute (Other); M.D. Anderson Cancer Center (Other); Phoenix Children's Hospital (Other); Alberta Children's Hospital (Other); University of Colorado, Denver (Other); Seattle Children's Hospital (Other); Johns Hopkins University (Other); Children's Mercy Hospital Kansas City (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-014
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Brain Cancer
Keywords: high-grade astrocytomas; newly diagnosed diffuse pontine tumors; External beam radiation therapy; cetuximab; irinotecan; POETIC
MeSH Terms: conditions — Brain Neoplasms | interventions — Cetuximab; Irinotecan

ARMS (2):
- pts with high-grade astrocytoma (Experimental): This is a 2-group parallel (high-grade astrocytoma, diffuse pontine tumor), single stage study investigating cetuximab in conjunction with external beam radiation therapy, followed by cetuximab and irinotecan in pediatric and young adult patients. Optional exploratory components of the study include (1) correlation of tumor molecular markers with outcome, (2) CSF proteomics, and (3) assay of serum cytokine levels in patients who develop a cetuximab-associated rash.
  Interventions: Other: cetuximab in conjunction with external beam radiation therapy, followed by cetuximab and irinotecan
- pts with diffuse pontine tumor (Experimental): This is a 2-group parallel (high-grade astrocytoma, diffuse pontine tumor), single stage study investigating cetuximab in conjunction with external beam radiation therapy, followed by cetuximab and irinotecan in pediatric and young adult patients. Optional exploratory components of the study include (1) correlation of tumor molecular markers with outcome, (2) CSF proteomics, and (3) assay of serum cytokine levels in patients who develop a cetuximab-associated rash.
  Interventions: Other: cetuximab in conjunction with external beam radiation therapy, followed by cetuximab and irinotecan

INTERVENTIONS:
Other: cetuximab in conjunction with external beam radiation therapy, followed by cetuximab and irinotecan — External beam radiation therapy (5940 cGy in 180 cGy fractions) with weekly cetuximab (250 mg/m2/dose).4-8 weeks rest, 10 cycles of irinotecan (16 mg/m2/day x 5 consecutive days x 2 weeks) with weekly cetuximab (250 mg/m2/dose) at about 21 day intervals. Research biological evaluations will be performed in consenting patients as an optional portion of the study. Cetuximab is to be given every 7 days (+/- 2 days). Cetuximab does not need to be given on Day 1 of each week.

SUMMARY:
Standard treatment for patients with diffuse pontine tumors is radiation therapy, but less than 10% of patients are cured. Adding standard chemotherapy has not improved the cure rate.

Standard treatment for high-grade astrocytomas is surgery and radiation. The surgeon removes as much of the tumor as she or he can. Radiation after that tries to kill any cancer cells that are left. Some patients also get chemotherapy. These are anti-cancer drugs. They can be given during or after radiation. Current standard treatments do not cure many patients.

In this study the doctors are adding a new medication called cetuximab to the treatment and will also use a chemotherapy medication (irinotecan) that has been promising for patients treated for recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either (1) histologic proof of a high-grade astrocytoma reviewed by a POETIC institutional pathologist or (2) a radiological diagnosis via MRI scan of a typical diffuse pontine tumor made by a POETIC institutional neuroradiologist. Patients with a radiological diagnosis via MRI scan of a typical diffuse pontine tumor will be enrolled on the diffuse pontine tumor arm of the study regardless of histology in cases that are biopsied. Note: For collaborating non-POETIC institutions, the reviews may be done by an institutional pathologist/neuroradiologist.
* Patients must begin study prescribed therapy within 42 days of neurosurgical resection or biopsy of the tumor (high-grade astrocytoma patients) or radiological diagnosis (diffuse pontine tumor patients).
* Age ≥ 3-years and < 22-years-old.
* Brain MRI (and any other studies done according to clinical indications) must not show any definitive evidence of leptomeningeal or extra-neural metastases.
* ANC ≥ 1000/μL and platelet count ≥ 100,000/μL
* Patients must have adequate organ function as defined by:
* Hepatic: total bilirubin < 1.5 mg/dl, AST ≤ 2.5 x the upper limit of normal.
* Renal: serum creatinine ≤ 1.5 x the upper limit of normal for age, or calculated creatinine clearance or nuclear GFR ≥ 70 ml/min/1.73 m2.
* The patient, or for minors, a parent or legal guardian, must give informed written consent indicating they are aware of the investigational nature of this study.

Exclusion Criteria:

* Evidence of leptomeningeal or extra-neural metastatic disease.
* Prior radiation therapy or chemotherapy
* Pregnancy, mothers unwilling to refrain from breast-feeding, and sexually mature patients unwilling to practice an effective form of birth control.
* Other significant concomitant medical illnesses that would compromise the patient's ability to receive all prescribed study therapy.
* Prior therapy which specifically and directly targets the EGFR pathway.
* Prior severe infusion reaction to a monoclonal antibody.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Patients with known Gilbert's Syndrome.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10-30 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (11):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - MD Anderson Cancer Center Orlando at Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - John Hopkins Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Md Anderson Cancer Center, Houston, Texas
  - Seattle Children'S Hospital, Seattle, Washington
- Alberta Children'S Hospital, Calgary, Alberta, Canada

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Started | 21 | 26
Completed | 20 | 25
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Full Range); unit: years] | 10.7 [3 to 19] | 6.4 [3 to 16] | 8.3 [3 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 4 | 6
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High-grade Astrocytoma and Diffuse Pontine Tumors Achieving One Year Progression Free Survival.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
Participants | 5 | 6

2. Primary Outcome: Number of Participants Experiencing Toxicity
Description: To determine the safety of cetuximab administered weekly in conjunction with involved field external beam radiation therapy for diffuse pontine tumors and high-grade astrocytomas, toxicities will be assessed via the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 3.0)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
Participants | 20 | 25

3. Secondary Outcome: Time to Progression
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
months | 9.02 [8.52 to 11.8] | 7.12 [6.89 to 12.5]

4. Secondary Outcome: Number of Participants Who Have Undergone Tumor Analysis
Description: Participant tumor analysis for potential associations between primary tumor tissue molecular markers and tumor response.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
Participants
  Tumor Analyzed | 18 | 1
  Tumor Did Not Undergo Analysis | 2 | 24

5. Secondary Outcome: Number of Samples Demonstrating EGFR Copy Number Gain
Description: Identify gene transcripts for putative cetuximab
Time Frame: 2 years
Population: Paraffin-embedded tumor sections were obtained from 19 of 23 patients who underwent surgery (18 HGA and one DIPG). Because only 1 DIPG sample was available and based on the number of available samples per arm it was pre-specified to pool data for this Outcome Measure.
Measure: Number; unit: samples
Groups:
- HGA and DIPG Tumors Analyzed: Paraffin-embedded tumor sections were obtained from 19 of 23 patients who underwent surgery (18 HGA and one DIPG tumors). Found tumor markers are reported as one group in the publication.
Arm/Group | HGA and DIPG Tumors Analyzed
Number analyzed (Participants) | 19
samples
  With GFR copy number gain | 18
  No GFR copy number gain | 1

6. Secondary Outcome: Number of Participant Tumors Analyzed for Potential Association Between Histology (Grade) With Protein and ELISA Measurements of Those Proteins.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
Participants
  Tumor tissue analysis completed | 18 | 1
  Tumor tissue analysis Not Done | 2 | 24

7. Secondary Outcome: Percentage of Participants With Development of Rash, Either Acneiform and/or Desquamation
Description: The purpose is to investigate whether the rash associated with cetuximab is secondary to an inflammatory pathway initiated and mediated by the action of cetuximab on host cells.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
percentage of participants | 60 | 53.3

8. Secondary Outcome: Event Free Survival
Time Frame: up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
months | 8.9 [5.8 to 11.8] | 6.9 [5.34 to 9.05]

9. Secondary Outcome: Overall Survival
Time Frame: Up to 43 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
Number analyzed (Participants) | 20 | 25
months | 17.4 [14.72 to 42.1] | 12.1 [9.93 to 18]

ADVERSE EVENTS:
Time Frame: Up to 43 months
Arm/Group | Pts With High-grade Astrocytoma | Pts With Diffuse Pontine Tumor
All-Cause Mortality (participants affected / at risk) | 16/21 | 24/26
Serious Adverse Events (participants affected / at risk) | 16/21 | 17/26
Other Adverse Events (participants affected / at risk) | 21/21 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With High-grade Astrocytoma (N=21) | Pts With Diffuse Pontine Tumor (N=26)
Ataxia (incoordination) (Nervous system disorders) | 0 | 1
CNS necrosis/cystic progression (Nervous system disorders) | 1 | 0
Colitis, infectious (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Extrpyrmdl/invlntry mvmnt/rstlssnss (Nervous system disorders) | 0 | 1
Hemorrhage, CNS (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 5 | 2
Hypotension (Vascular disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Inf norm ANC/gr1/2 neut-Blood (Infections and infestations) | 0 | 1
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Infections and infestations) | 1 | 0
Inf unknown ANC-Blood (Infections and infestations) | 0 | 1
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 0 | 1
Infection, other (Infections and infestations) | 3 | 3
Intra-operat injury- Brain (Injury, poisoning and procedural complications) | 0 | 1
Keratitis (corneal inflamm/ulceratn) (Eye disorders) | 0 | 2
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 1 | 0
Lymphopenia (Investigations) | 0 | 3
Mood alteration - Agitation (Psychiatric disorders) | 0 | 1
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Neurology - Other (specify) (Nervous system disorders) | 1 | 1
Neuropathy: cranial - CN II Vision (Nervous system disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 2 | 2
Nrpthy:cranl-CN IX Mtr-phrynx;snsry-ear,phrynx,tng (Nervous system disorders) | 1 | 0
Nrpthy:cranl-CN X Mtr-palate;phrynx,lrynx (Nervous system disorders) | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 | 0
Pain - Head/headache (Nervous system disorders) | 2 | 1
Pain - Pain NOS (General disorders) | 1 | 0
Personality/behavioral (Psychiatric disorders) | 1 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 3
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Renal/Genitourinary-Other Specify (Renal and urinary disorders) | 1 | 0
Seizure (Nervous system disorders) | 4 | 2
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1
Somnolence/dprssd level of conscious (Nervous system disorders) | 0 | 1
Speech impairment (Nervous system disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
Urinary retention (includ neurogenic bladder) (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Weight loss (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With High-grade Astrocytoma (N=21) | Pts With Diffuse Pontine Tumor (N=26)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 | 7
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 2 | 0
ALT, SGPT (Investigations) | 9 | 5
Anorexia (Metabolism and nutrition disorders) | 9 | 10
AST, SGOT (Investigations) | 6 | 4
Ataxia (incoordination) (Nervous system disorders) | 5 | 11
Auditory/Ear, other (Ear and labyrinth disorders) | 0 | 3
Bicarbonate, serum-low (Investigations) | 3 | 0
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 3 | 7
Cushingoid appearance (Endocrine disorders) | 2 | 11
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 5
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 7 | 9
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 | 3
Dizziness (Nervous system disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 0 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Fever (in the absence of neutropenia) (General disorders) | 3 | 3
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 5
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 3
Hearing:pts w/o BL audiogm & not enroll in mon prg (Ear and labyrinth disorders) | 0 | 2
Hemoglobin (Blood and lymphatic system disorders) | 6 | 5
Hydrocephalus (Nervous system disorders) | 7 | 3
Hypotension (Vascular disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Incontinence, urinary (Renal and urinary disorders) | 0 | 3
Inf norm ANC/gr1/2 neut-Mucosa (Infections and infestations) | 0 | 3
Inf norm ANC/gr1/2 neut-Myositis infection(muscle) (Infections and infestations) | 0 | 2
Inf norm ANC/gr1/2 neut-Otitis externa (Infections and infestations) | 2 | 0
Inf unknown ANC-Cellulitis(skin) (Infections and infestations) | 0 | 4
Infection, other (Infections and infestations) | 8 | 11
Intra-op injury- CN VII (facial) motor-face (Injury, poisoning and procedural complications) | 0 | 2
Keratitis (corneal inflamm/ulceratn) (Eye disorders) | 0 | 2
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 2 | 0
Leukocytes (total WBC) (Investigations) | 9 | 13
Lymphopenia (Investigations) | 15 | 20
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Mood alteration - Agitation (Psychiatric disorders) | 2 | 3
Mood alteration - Anxiety (Psychiatric disorders) | 0 | 4
Muscle weakness - Left-sided (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness - Right-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 10 | 7
Neurology - Other (specify) (Nervous system disorders) | 6 | 2
Neuropathy: motor (Nervous system disorders) | 6 | 13
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 | 11
Nrpthy:cranl-CN III Pupl,upp eyeld, extrclr mvmnts (Nervous system disorders) | 0 | 3
Nrpthy:cranl-CN IV Dwnwrd,inwrd eye mvmnt (Nervous system disorders) | 0 | 2
Nrpthy:cranl-CN IX Mtr-phrynx;snsry-ear,phrynx,tng (Nervous system disorders) | 0 | 4
Nrpthy:cranl-CN VI Ltrl eye dviatn (Nervous system disorders) | 0 | 10
Nrpthy:cranl-CN VII Mtr-face;snsry-taste (Nervous system disorders) | 3 | 5
Nrpthy:cranl-CN VIII Hearing,balance (Nervous system disorders) | 0 | 2
Nrpthy:cranl-CN X Mtr-palate;phrynx,lrynx (Nervous system disorders) | 0 | 6
Nrpthy:cranl-CN XI Mtr-strnmstd,trpzius (Nervous system disorders) | 2 | 0
Nrpthy:cranl-CN XII Motor-tongue (Nervous system disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 2 | 0
Ocular surface disease (Eye disorders) | 0 | 3
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2 | 0
Otitis, external ear (non-infect) (Ear and labyrinth disorders) | 0 | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 6
Pain - Head/headache (Nervous system disorders) | 10 | 8
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 | 0
Platelets (Investigations) | 2 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 10 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 0
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyramidal tract dysfunction (Nervous system disorders) | 2 | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 9
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 7 | 7
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 0
Seizure (Nervous system disorders) | 6 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 2
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 4
Somnolence/dprssd level of conscious (Nervous system disorders) | 2 | 3
Speech impairment (Nervous system disorders) | 2 | 6
Supraventricular arrhythmia NOS (Cardiac disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Vision-blurred vision (Eye disorders) | 0 | 2
Voice changes/dysarthria (Nervous system disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 13 | 12
Weight gain (Investigations) | 5 | 3
Weight loss (Investigations) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT01012609/Prot_SAP_000.pdf